CLINICAL TRIAL: NCT00670215
Title: Prospective, Randomized, Double-blind, Comparison of Ciprofloxacin Extended-release 1000 mg Tablets Given as Two Different Prophylactic Dosing Regimens (Regimen I - Single-dose Ciprofloxacin MR 1000 mg or Regimen II - Multiple-dose Ciprofloxacin MR 1000 mg Once Daily for 3 Days) for the Prevention of Post-operative Infectious Complications in Patients Undergoing Transrectal Needle Biopsy of the Prostate
Brief Title: BAYQ3939, 1000 mg Tablet in Transrectal Needle Biopsies of the Prostate (TRNBP) - Infection Prophylaxis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 100588
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Bacterial Infections
Keywords: Prevention of infectious complications; transrectal needle biopsies of the prostate; TRNBP
MeSH Terms: conditions — Bacterial Infections | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Ciprofloxacin single dose
- Arm 2 (Experimental)
  Interventions: Drug: Ciprofloxacin triple dose

INTERVENTIONS:
Drug: Ciprofloxacin single dose — Patients randomized to this regimen will receive a single-dose of ciprofloxacin MR 1000 mg PO approximately 2 to 3 hours prior to the TRNBP. Patients will also receive two doses of matching placebo approximately 24 hours prior to and approximately 24 hours after the TRNBP.
  Arms: Arm 1
Drug: Ciprofloxacin triple dose — Patients randomized to this regimen will receive three doses of ciprofloxacin MR 1000 mg PO. The doses will be approximately 24 hours prior to the TRNBP, approximately 2 to 3 hours prior to the TRNBP, and approximately 24 hours after the TRNBP.
  Arms: Arm 2

SUMMARY:
The primary purpose of this clinical trial is to compare in a double-blind randomized trial, the efficacy and safety of ciprofloxacin MR 1000 mg tablets given as a single-dose or as a multiple-dose regimen for the prevention of infectious complications in patients undergoing transrectal needle biopsies of the prostate (TRNBP).

ELIGIBILITY:
Inclusion Criteria:

* Transrectal needle biopsy of the prostate required.
* A clean-catch midstream-urine (MSU) culture negative (<104 CFU/mL) for possible pathogens at the Pre-Therapy Visit prior to the TRNBP.
* Gastrointestinal absorption is adequate as evidenced by passage of gas or feces per rectum and patient can tolerate oral food, fluids, and medication without vomiting or diarrhea.

Exclusion Criteria:

* History of hypersensitivity to ciprofloxacin or other quinolone antibiotics
* Valvular heart disease that requires antibiotic prophylaxis to prevent bacterial endocarditis
* Concomitant use of theophylline, probenecid, or warfarin at any time during the entire study
* Renal insufficiency
* Known or suspected central nervous system disorder that may predispose to seizures or lower the seizure threshold
* Absolute neutrophil count (ANC) <1000/mm3
* Human immunodeficiency virus (HIV) infection with a CD4 count <200 cells/micL. HIV testing is NOT required
* Antibiotic administration within one week of the TRNBP
* Severe hepatic insufficiency (Child-Pugh C)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2004-04; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Bacteriological Response (bacteriuria vs. no bacteriuria) | 10-14 days after last dose of study med

SECONDARY OUTCOMES:
Clinical Response (patients without clinical symptoms or signs of bacteriuria vs. patients with clinical symptoms or signs of bacteriuria) | 10-14 days after last dose of study med.
Incidence of post-procedure GU tract infections other than bacteriuria | any time after the TRNBP

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (50):
- United States (18):
  - Birmingham, Alabama
  - San Diego, California
  - San Francisco, California
  - Sherman Oaks, California
  - Waterbury, Connecticut
  - Ocala, Florida
  - Atlanta, Georgia
  - Roswell, Georgia
  - Chicago, Illinois
  - Hopedale, Massachusetts
  - New Brunswick, New Jersey
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Simpsonville, South Carolina
  - San Antonio, Texas
  - Norfolk, Virginia
  - Spokane, Washington
- Brazil (5):
  - Salvador, Estado de Bahia
  - Belo Horizonte, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
  - Rio de Janeiro
- Canada (11):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Victoria, British Columbia
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Fleurimont, Quebec
  - Laval, Quebec
  - Québec, Quebec
- Italy (5):
  - Bergamo
  - Milan
  - Napoli
  - Padua
  - Roma
- Mexico (6):
  - Zapopan, Jalisco
  - México D.F., Mexico
  - Villahermosa, Tabasco
  - México, D. F.
  - México, D.F.
  - Monterrey
- Spain (5):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Vigo, Pontevedra
  - Seville, Sevilla
  - Valencia, Valencia